CLINICAL TRIAL: NCT06833788
Title: Treatment of Anaemia After Caesarean With Intravenous Versus Oral Iron and Postpartum Depression: a Multicentric Randomized Open-labelled Controlled Trial
Brief Title: Treatment of Anaemia After Caesarean With Intravenous Versus Oral Iron and Postpartum Depression
Acronym: IRON-DEP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: APHP220806; 2023-503283-17-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Postpartum Depression (PPD)
Keywords: Postpartum depression (PPD); Postpartum anaemia; Caesarean; Intravenous (IV) iron therapy; Oral iron therapy
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous iron (Experimental): Women in the experimental arm will receive an IV iron infusion within 5 days after delivery
- Oral iron (Active Comparator): Women in the comparator arm will receive oral iron supplementation for 8 weeks after delivery

INTERVENTIONS:
Drug: Ferric carboxymaltose IV — Single dose of Ferric carboxymaltose 1000 mg (20mL) IV infusion (20ml vial of 1000mg iron or two 10ml vials of 500mg)
Drug: TIMOFÉROL® — 100 mg once a day (2 pills of TIMOFÉROL® 50mg)

SUMMARY:
The objectif of the IRON-DEP Study is to assess the efficacy of intravenous (IV) versus oral iron treatment on the prevalence of postpartum depression (PPD) in women with moderate iron deficiency anemia after caesarean delivery.

DETAILED DESCRIPTION:
PPD is a frequent (10-20% of delivery) and serious condition that has a detrimental impact on both maternal and child health by altering the quality of their interactions. Moreover, it is a significant risk factor for suicide, which is the leading cause of maternal death.

The increased risk of PPD in women with postpartum anemia has been documented. Women who delivered by cesarean are particularly vulnerable to this risk as this mode of delivery is a risk factor for both postpartum anaemia and postpartum depression. Therefore, correcting anemia and preventing PPD in this population represent a major public health priority.

First line treatment recommended for iron deficiency moderate anaemia (8.0g/dL≤ Hb ≤10.0g/dL) is oral iron. However oral iron is associated with very frequent adverse effects, contributing to poor tolerance and compliance of this treatment. Actually, IV iron is indicated in women with non-severe postpartum anaemia with lack of response or intolerance to oral iron treatment. There is growing interest in the use of intravenous iron and several randomized controlled trials demonstrated that IV iron is significantly more efficient than oral iron supplementation to correct moderate postpartum anaemia and increase haemoglobin level. However, none of them compared the efficacy of IV iron versus oral iron on postpartum depression as a primary outcome.

The hypothesis of the IRON-DEP Study is that, among women with moderate postpartum iron deficiency anaemia after caesarean delivery, the prevalence of PPD symptoms at 8 weeks after delivery is lower in women treated with IV iron than in those treated with oral iron.

The IRON-DEP trial is a phase IV national multicenter comparative randomized controlled superiority open-label trial with 2 parallel groups.

Implementation of the study :

* 24 french maternity units will be participating
* Women who delivered by cesarean admitted in the postpartum maternity ward, with postpartum anaemia will be screened to check the inclusion and exclusion criteria.
* The investigator will inform the eligible patient about the protocol and obtain the written consent
* The randomization will take place during the hospitalization for caesarean delivery and will be stratified on the centre and on the initial severity of post-partum anemia (according to the postpartum hemoglobin level).
* IV iron will be administered during hospitalization and participants in the oral iron group will start their treatment during their hospitalization for 8 weeks treatment.
* A follow up visit at 8 weeks postpartum will be planned at the maternity unit for all participants
* All participants will fill in self-assessment questionnaires (online or paper form) at inclusion, 8 weeks and 6 months postpartum follow up.

ELIGIBILITY:
Pre-inclusion criteria:

* Age ≥18 years
* Caesarean delivery (elective or in emergency)
* Gestational age at delivery ≥ 32 weeks
* 8.0 g/dL ≤ postoperative Hb level ≤ 10.0 g/dL measured within 72 hours postpartum
* Informed consent form signed
* Hospitalization in the postpartum maternity ward
* National social security coverage including AME

Inclusion criteria:

* Ferritinemia ≤ 100 ng/mL OR transferrin saturation ≤ 20% measured after postoperative Hb level measurement
* EPDS score in the immediate postpartum <11 with a "never" answer to question n°10

Exclusion Criteria:

* Stillbirth or neonatal death
* Body weight < 35kg or > 100kg at the end of pregnancy
* Biermer disease
* Hemochromatosis
* Homozygous sickle cell disease or thalassemia
* Chronic iron supplementation (outside pregnancy)
* Known hypersensitivity or allergy to the studied drugs (IV or oral iron)
* Contra-indication to the studied drugs (IV or oral iron)
* Severe asthma (with daily background treatment)
* Any known severe renal or liver disorder
* Active acute infection
* Diagnosis of schizophrenia or physical and intellectual state incompatible with a reliable self-evaluation
* Women currently treated with medication or with Electro Convulsion Therapy (ECT) for depression or bipolar disorders
* Participation in another clinical trial involving an intervention with the following risks:

  * A change (increase or decrease in value) in Haemoglobin measured at 2 months postpartum OR
  * A change in EPDS score measured at 2 and 6 months postpartum OR
  * A trial exploring an intervention with a specific anaphylactic risk (reported as a potential adverse events in the protocol of the other trial) administered during the postpartum hospitalization period.
* Poor understanding of the French language
* Legal protection (curatorship or tutorship)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2860 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of PostPartum Depression (PPD) symptoms defined by an Edinburg Postpartum Depression Scale (EPDS) score ≥ 11 | 8 weeks postpartum
  Edinburg Postpartum Depression Scale (EPDS) wil be measured by a self-assessment questionnaire at 8 weeks.
  The primary measure of treatment effect will be based on the 'treatment policy' estimand: the effect will be measured by including all women who participated in the study, according to the initial randomization, regardless of the treatment they actually received or their adherence to the treatment. If the 8-week value is not observed, these participants will be included in the analysis after imputing their missing value.
  Secondary measures of treatment effect will be implemented based on the "principal stratum strategy" estimand: the effect will be measured in women according to the treatment they actually received and in those who achieved a compliance rate of over 80%.
  The estimands discussed above will be applied to all efficacy-related criteria. For safety-related criteria, only the second estimand (principal stratum strategy) will be considered.

SECONDARY OUTCOMES:
The mean Haemoglobin (Hb) level | 8 weeks postpartum
  All participants will have à haemoglobin measurment at 8 weeks
Change in postpartum Haemoglobin (Hb) level | At Inclusion and at 8 weeks postpartum
  Haemoglobin measurment at 8 weeks
The proportion of women with Haemoglobin level < 12.0 g/dL | 8 weeks postpartum
  Haemoglobin measurment at 8 weeks
The mean ferritinemia level | At Inclusion and at 8 weeks postpartum
  Ferritinemia dosage at 8 weeks
The mean change in ferritinemia level | At Inclusion and at 8 weeks postpartum
  Ferritinemia dosage at 8 weeks
The proportion of women with ferritinemia < 20 ng/mL | 8 weeks postpartum
  Ferritinemia dosage at 8 weeks
Mean EPDS score | 8 weeks postpartum, 6 months postpartum
  Edinburg Postpartum Depression Scale (EPDS) wil be measured by a self-assessment questionnaire
The proportions of participants with moderate depressive symptoms level defined by an EPDS ≥ 11 and <13 | 8 weeks postpartum, 6 months postpartum
  Edinburg Postpartum Depression Scale (EPDS) will be measured by a self-assessment questionnaire
The proportions of participants with high depressive symptoms level defined by an EPDS ≥13 | 8 weeks postpartum, 6 months postpartum
  Edinburg Postpartum Depression Scale (EPDS) wil be measured by a self-assessment questionnaire
The mean change in EPDS score | 8 weeks postpartum, 6 months postpartum
  Edinburg Postpartum Depression Scale (EPDS) wil be measured by a self-assessment questionnaire
The need for red blood cell transfusion | From discharge to 8 weeks postpartum
  The variable of interest is whether (yes or no) a patient received a red blood cell transfusion. The summary measure of the effect is the percentage of patients who were transfused.
The mean fatigue score measured by the Multidimensional Fatigue Inventory score-20 (MFI-20) | 8 weeks postpartum, 6 months postpartum
  Multidimensional Fatigue Inventory score-20 (MFI-20) self-assessment questionnaire ( overall and in each of its 5 dimensions: general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue).
The proportion of women with high fatigue score (MIF-20 score>15) | 8 weeks postpartum, 6 months postpartum
  Multidimensional Fatigue Inventory score-20 (MFI-20) self-assessment questionnaire
The mean relative change in MFI-20 scores | 8 weeks postpartum, 6 months postpartum
  Multidimensional Fatigue Inventory score-20 (MFI-20) self-assessment questionnaire
The mean score for mother and child bonding measured by the Mother to Infant Bonding Scale (MIBS) | 8 weeks postpartum, 6 months postpartum
  Mother to Infant Bonding Scale (MIBS) self-assessment questionnaire
The proportion of women with MIBS≥2 | 8 weeks postpartum, 6 months postpartum
  Mother to Infant Bonding Scale (MIBS) self-assessment questionnaire
The proportion of breastfeeding women and mean duration for those who stopped | 8 weeks postpartum, 6 months postpartum
  Participants will answer self assessment questionnaires
The mean relative change in MIBS score | 8 weeks postpartum, 6 months postpartum
  Mother to Infant Bonding Scale (MIBS) self-assessment questionnaire
The mean score of quality of life measured by EQ-5D-5L (European questionnaire of quality of life, 5 domains, 5 levels) | 8 weeks postpartum, 6 months postpartum
  EQ-5D-5L (European questionnaire of quality of life, 5 domains, 5 levels) overall and for each of the 5 dimensions
The number of women in each group who also received the other group treatment within 8 weeks postpartum | Up to 8 weeks
  Women who needed IV iron in the oral iron group because of poorly tolerated anaemia, and women who took oral iron after hospital discharge in the IV iron group
Assessement of adverse events | From first drug administration to 8 weeks
  Incidence, nature, and severity of adverse events and serious adverse events
Compliance to treatment for participants in the oral iron arm | 8 weeks
  Good compliance defined by the overall drug intake >80% of the prescribed oral iron treatment
Total costs of healthcare resources for medicoeconomic cost-consequence analysis | Up to 6 months postpartum
  Use of resources and consequences for women are collected prospectively from the time of randomization up to 6 months by a a self-assessment questionnaire at 8 weeks and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre BONNET, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris; Catherine DENEUX-THARAUX, MD, PhD, Study Director — Assistance Publique Hopitaux de Paris
Locations (1):
- CHU Armand -Trousseau, AP-HP Service d'anesthésie-réanimation chirurgicale, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF